CLINICAL TRIAL: NCT06013878
Title: Biomechanical Validation of the Caregiver Assisted Transfer Technique Instrument
Brief Title: Biomechanical Validation of the CATT
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F4539-R; 1I01RX004539-01A1 (NIH)
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Informal Caregivers; Low Back Pain; Biomechanics
Keywords: caregivers; outcome assessment, health care; wheelchairs; physical medicine and rehabilitation; moving and lifting patients
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Informal Caregivers: Informal caregivers who provide transfer assistance to an individual with a disability
  Interventions: Other: Transfer Training with clinician
- Individuals who use transfer assistance: Individuals who require assistance with transfers moving from one surface to the other
  Interventions: Other: Transfer Training with clinician

INTERVENTIONS:
Other: Transfer Training with clinician — Participants will undergo transfer training with a clinician who is an expert on assisted transfer techniques if they are found to have skill deficits during the study. After training, a transfer assessment will be conducted to examine if the transfer skills of the caregiver have improved

SUMMARY:
As of 2020, 53 million Americans provide unpaid care to an individual with a disability. One commonly performed activity of daily living (ADL) provided by informal caregivers is assisted transfers, which requires moving an individual from one surface to another. Approximately 94% of informal caregivers who assist with ADLs to persons with adult-onset chronic physical disabilities affecting mobility reported musculoskeletal discomfort, with pain and discomfort made worse by performing caregiving activities. Although many informal caregivers assist with transfers, most have never received any formal training in proper manual lifting or mechanical lifting techniques. Improper transfer techniques can be detrimental to not only caregiver health but also to the persons they assist resulting in shoulder injury, bruising and pain from manual lift techniques, hip fractures from falls, and skin tears from shear force that occurs with sliding during transfers. Current standard of care provides limited in-person training of caregivers, as most of the rehabilitation process is client-focused. When training is provided clinicians have no means to objectively evaluate if proper techniques are being performed at discharge or when the caregiver and care recipient return home. For this reason, an outcome measure called the Caregiver Assisted Transfer Technique Instrument (CATT) was developed to provide a quick, objective way to evaluate proper technique of caregivers who provide transfer assistance to individuals with disabilities. The CATT evaluates the caregiver's performance on setup, quality of the task performance, and results. After a formal assessment through stakeholder review involving clinicians, informal caregivers, and individuals with physical disabilities who require transfer assistance, the CATT was expanded to include two versions; one that evaluates manual lift technique (CATT-M) and one that evaluates mechanical lift techniques (CATT-L). However, the CATT must undergo further testing with informal caregivers and the individuals they assist to determine if the CATT is a reliable, valid, and responsive tool for identifying skill deficits in caregivers performing assisted transfers. The purpose of this study is to establish the psychometric properties (reliability, validity, and responsiveness) of the CATT and to evaluate the effects of an individualized training session for participants who have transfer technique deficits as identified by the CATT. The long-term goal of this research is to develop the CATT so that it can be used as an objective indicator of transfer performance as well as guide training and educational interventions for informal caregivers to reduce the risk of musculoskeletal pain and injury associated with assisted transfers.

DETAILED DESCRIPTION:
The objective of this study is to further establish the psychometric properties of the CATT and to evaluate the effects of an individualized intervention for participants who have transfer technique deficits as identified by the CATT.

Specific Aim 1 (Reliability): Establish the CATT's intra and inter-rater reliability in evaluating the quality of informal caregiver assisted transfer techniques.

Hypothesis 1a: Each item and the total score of the CATT will have excellent intra-rater and interrater reliability (ICC >0.8 for total scores; K>0.8 for individual item scores).

Specific Aim 2 (Validity): Establish the CATT's construct and concurrent validity through relating the scores to caregiver characteristics and to the biomechanical measurement of caregiver techniques.

Hypothesis 2a (Construct Validity): Characteristics of the caregiver including younger age, lower levels of shoulder, neck or back pain, better overall health status, higher income, and higher level of education will predict higher scores on the CATT (indicative of better transfer technique).

Hypothesis 2b (Concurrent Validity): Higher total CATT scores (indicative of better transfer technique) will correlate with lower peak lumbar forces, less trunk flexion and axial rotation, and greater hip and knee flexion.

Specific Aim 3 (Responsiveness): Demonstrate improvement in the quality of assisted transfer technique after individualized training with caregivers who have transfer skill deficits.

Hypothesis 3a: After training, participants will demonstrate higher CATT scores, showing improvement in transfer technique.

Hypothesis 3b: After training, the biomechanical measures described in Specific Aim 2 will show improvement (e.g., lower peak lumbar forces, less trunk flexion and axial rotation, and greater hip and knee flexion).

This study (observational cohort study) will be conducted with a convenience sample of informal caregivers and their care recipients who they transfer. After signing informed consent, all participants will complete a series of baseline questionnaires consisting of their demographic information, health status, quality of life, and pain. After completion of the surveys, several anthropometric measurements of the caregiver will be taken by the research team, including height, weight, length of the foot, shank, thigh, and trunk. Caregiver participants will then be fitted with eight wireless inertial measurement units placed on the their feet, legs, and trunk. They will also be fitted with pressure insoles placed on the inside of their shoes.

Participants will be asked to perform transfers from the wheelchair to two surfaces that they normally transfer to during daily living. A variety of surfaces will be made available for participants to transfer, including a bench, a mat table, a commode, a bed, a chair, a wheelchair and a recreational mobility device (hand cycle). Additional surfaces may be provided at the participant's request. If pairs normally use a transfer assist device to facilitate the transfer, assistive technologies will be made available to them so they can complete the transfers in their usual manner (transfer boards and mechanical lifts will be available on site). The participants will be asked to perform four transfers: 1) moving from the wheelchair to the first selected surface, 2) moving from the first selected surface back to their wheelchair, 3) moving from the wheelchair to the second selected surface and 4) moving from the second selected surface back to the wheelchair. During each transfer, three expert raters will watch each transfer and score the version of the CATT that corresponds with the caregiver's transfer method. Participant dyads will be asked to return to the lab, or the research team will return to them between 24 and 72 hours later to perform the transfer portion of the protocol again. This time frame helps to ensure that repeat administration of the CATT is not affected by rater memories of the first assessment. All raters will independently score each complete and incomplete transfer using the CATT. Raters will also be asked to score the video recordings of the transfers at a later date (at least 1 week after the live recordings).

Outcome measures including surveys, questionnaires, and CATT scores from raters will be collected and managed using an online survey approved by the VA Pittsburgh Healthcare System. During the transfers, three rehabilitation professionals will rate each transfer using the CATT while biomechanical data are collected using a combined IMU/pressure insole system. A webcam integrated into the Ultium IMU/insole system will also record each transfer to facilitate determination of the specific phases of the transfer process.

Participants who were identified as having transfer skill deficits (i.e. scoring a zero on at least two CATT items) in Visit 1 will be asked to participate in a training session during Visit 2 to determine the responsiveness of a CATT-based training protocol. A clinician trained on the CATT will conduct the training session. The clinician will work with the participants to learn and practice the new techniques. They will have an opportunity to practice the techniques until they feel comfortable with performing them. They will be asked to perform a minimum of two transfers to the same surface for the reassessment. A rater who is trained on the CATT but blinded to the biomechanical deficits and training intervention will score the participants using the CATT after training.

ELIGIBILITY:
Inclusion Criteria:

Individuals who use assistance with transfers and their caregivers will be recruited for this study.

Caregiver participants will be included in the study if they meet the following criteria:

1. at least 18 years old
2. routinely provide transfer assistance to an adult with a physical disability
3. serving as a caregiver for at least 3 months
4. no formal didactic or structured training on assisted transfer techniques received as part of a professional degree or training program

Care recipient participants will be included in the study if they meet the following criteria:

1. at least 18 years old,
2. has a physical disability diagnosis for at least one year
3. requires assistance with transfers
4. currently receives care from an informal caregiver

Exclusion Criteria:

Caregiver participants will be excluded if they:

1) have a current or recent history of back, neck, or other type of musculoskeletal injury within the last 6 months that would be exacerbated by performing an assisted transfer

Care recipient participants will be excluded if they:

1. have existing pressure ulcers or a recent history of pressure ulcers within the last 3 months
2. have any recent upper extremity injuries (within the last 6 months) that could be exacerbated by being transferred

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caregivers and care recipients who are eligible for the study will be recruited through community locations, including rehabilitation facilities, organizations that provide services to both caregivers and individuals with physical disabilities, research registries for individuals with disabilities, and at at national and local rehabilitation events, disability conferences and expos.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Caregiver Assisted Transfer Technique Instrument (CATT) Scores | Change from baseline and after intervention at 1 week
  An outcome measure called the Caregiver Assisted Transfer Technique Instrument (CATT) was developed to provide a quick, objective way to evaluate proper technique of caregivers who provide transfer assistance to individuals with disabilities. The CATT consists of two versions; one that evaluates manual lift technique (CATT-M) and one that evaluates mechanical lift techniques (CATT-L). It uses three subdomains (set up, transfer performance, and results) to assess caregiver technique during transfers. The investigators expect to see improvements in CATT Scores (higher scores) after intervention with a therapist.

SECONDARY OUTCOMES:
Change in peak lumbar extension moments | Change from baseline and after intervention at 1 week
  High lumbar extension moments have been associated with poor lifting technique. Using proper lifting technique has been shown to reduce moments at the L5/S1 joint. The investigators expect to see lower lumbar extension moments after a transfer training intervention with a therapist. Lumbar extension moments will be determined using an inverse dynamics model with data from IMUs and pressure insoles as inputs to the model.
Change in peak lumbar compression forces | Change from baseline and after intervention at 1 week
  High Lumbar compression forces at L5/S1 have been associated with low back pain in caregivers who perform lifting tasks. Using proper lifting techniques have been shown to reduce compressive forces at the L5/S1 joint. The investigators expect to see lower lumbar compressive forces after transfer training with a therapist. Lumbar compressive forces will be determined using an inverse dynamics model, with raw data from IMUs and pressure insoles at the model inputs.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia M Koontz, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No